CLINICAL TRIAL: NCT03490097
Title: Benefits of Statins in Chronic Hepatitis C Patients Receiving Sofosbuvir/Daclatasvir Combination
Brief Title: Statins in Chronic Hepatitis C Patients Receiving Sofosbuvir/Daclatasvir Combination
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Mahmoud Shaheen, Associate Professor, Faculty of pharmacy, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHCL35
Record Dates: First submitted 2018-03-19; First posted 2018-04-06 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Chronic Hepatitis c; Metabolic Syndrome
MeSH Terms: conditions — Hepatitis C, Chronic; Metabolic Syndrome | interventions — Simvastatin; Sofosbuvir; daclatasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Experimental): low dose of simvastatin10 mg plus sofosbuvir 400mg / daclatasvir 60 mg daily for 12 weeks.
  Interventions: Drug: Simvastatin 10mg; Drug: sofosbuvir plus daclatasvir
- Group II (Active Comparator): sofosbuvir plus daclatasvir
  Interventions: Drug: sofosbuvir plus daclatasvir

INTERVENTIONS:
Drug: Simvastatin 10mg — tablets
  Other Names: simvastatin
  Arms: Group I
Drug: sofosbuvir plus daclatasvir — sofosbuvir 400mg daclatasvir 60 mg daily for 12 weeks.
  Other Names: Sovodac

SUMMARY:
The purpose of the study is to determine if statin can affect the clinical outcome of chronic hepatitis C patients receiving Sofosbuvir/Daclatasvir/Ribavirin combination

DETAILED DESCRIPTION:
Aim of the work

To determine the benefits of statin use in CHC patients treated with Sofosbuvir/Daclatasvir/Ribavirin through :

Primary Outcome: Assessment of therapeutic SVR12

Seconadry Outcome

1. assessment of Chronic hepatitis C(CHC) infection risk on development of metabolic syndrome through assessment of lipid profile , fasting glucose test , HgbA1C and C-reactive protein(CRP).

2- Evaluation of CHC related complications such as fibrosis and cirrhosis

Patients will be followed up for the whole study period and will be subjected to assessment of the following:

1. CBC , liver function test , lipid profile and CK every month till the end of therapy.
2. HgA1C and CRP at the end of therapy.
3. HCV-PCR test 3 months after the end of therapy.
4. Fibrosis using (FIB-4) 3 months after the end of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients age 18 to 70 years old.
2. Easy to treat group: treatment naïve patients with serum HCV RNA positivity by PCR.
3. Clinically stable condition outpatients.
4. Platelet count ≥ 150,000/mm³.
5. INR ≤ 1.2.
6. Serum albumin ≥ 3.5 g/dl.
7. Total serum bilirubin ≤ 1.2 mg/dl.

Exclusion Criteria:

1. Inadequately controlled diabetes mellitus (HbA1c > 9%) .
2. Total serum bilirubin > 3mg/dl.
3. HCV-HIV co infection.
4. HBV-HCV co infection.
5. Any cause for chronic liver disease other than hepatitis C
6. Uncontrolled hypothyroidism.
7. Hepatocellular carcinoma, except 4 weeks after intervention aiming at cure with no evidence of activity by dynamic imaging (CT or MRI).
8. Extra-hepatic malignancy except after two years of disease-free interval.
9. Child's C cirrhotic patients.
10. Creatinine kinase > 350 u/l

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
SVR 12 | 3 months after end of therapy
  sustained virological response 3 months after the end of therapy

SECONDARY OUTCOMES:
Lipid marker | three months
  lipid profile
Glycemic status marker | three months
  fasting glucose test
inflammatory marker | three months
  C-reactive protein(CRP).

OTHER OUTCOMES:
CHC related complications | 6 months
  fibrosis and cirrhosis

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Ali Sabri, Professor, Study Director — Professor of clinical pharmacy , ASU
Locations (1):
- Kobri El koba Armed Forces Hospital, Cairo, Egypt